CLINICAL TRIAL: NCT07024277
Title: A Phase II Study Evaluating the Preliminary Efficacy and Safety of ZG006 in Participants With Metastatic Neuroendocrine Prostate Cancer
Brief Title: Study of ZG006 in Participants With Neuroendocrine Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-005
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Neuroendocrine Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part2 (Experimental): Participants will receive the RP2D identified in Part 1 of the study.
  Interventions: Biological: ZG006
- Part 1 (Experimental): The preliminary efficacy and safety of ZG006 at the two determined potential Phase II recommended doses (10 mg and 30 mg) will be assessed in Participants with advanced metastatic NEPC.
  Interventions: Biological: ZG006

INTERVENTIONS:
Biological: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.

SUMMARY:
This is a multicenter, open-label Phase II study, aimed at exploring the preliminary efficacy and safety of ZG006 in patients with advanced metastatic NEPC who have previously failed standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male Participants aged 18 to 80 years (inclusive);
* Advanced metastatic neuroendocrine prostate cancer;
* disease progression after at least one line of platinum-based systemic therapy or intolerance to toxicity;
* Measurable disease according to RECIST v1.1 criteria;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* Known positive test for human immunodeficiency virus (HIV) or hepatitis；
* Patients were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Modified Best Overall Response（mBOR） | Baseline to 12 months
  mBOR will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 with Prostate Cancer Working Group 3 (PCWG3) modifications.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Baseline to 12 months
Overall Survival (OS) | Baseline to 12 months
Disease Control Rate (DCR) | Baseline to 12 months
Adverse Events（AE） | Day 1 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Fudan university shanghai cancer center, Shanghai, Shanghai Municipality, China